CLINICAL TRIAL: NCT06200922
Title: Telehealth in the Rehabilitation of Urinary Incontinence in Older Women: Randomized Controlled Trial
Brief Title: Telehealth in the Rehabilitation of Urinary Incontinence in Older Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Luis Henrique Telles da Rosa, Clinical Professor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFCSPAUI
Record Dates: First submitted 2023-11-14; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Urinary Incontinence in Old Age
Keywords: Urinary Incontinence; Old Age; Pelvic Physiotherapy; Telehealth; Telerehabilitation
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Participants will be divided into three groups: Synchronous Group: will receive guidance and perform a real-time guided pelvic physiotherapy protocol through online physiotherapy by the physiotherapist, Asynchronous Group: will receive guidance and perform a pelvic physiotherapy protocol after the evaluation, without the real-time monitoring by the physical therapist and face-to-face group: will receive guidelines and will perform a pelvic physiotherapy protocol oriented in person by the physical therapist. All groups will receive the same treatment for 12 weeks, which will include floor muscle training pelvic floor, urge suppression techniques, bladder training and behavioral therapy.
Who Masked: Outcomes Assessor
Masking Description: The evaluations will be performed by a different researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Synchronous Group (Experimental): Will receive guidance and perform a real-time guided pelvic physiotherapy protocol through online physiotherapy by the physiotherapist.
  Interventions: Other: Pelvic physiotherapy
- Asynchronous Group (Experimental): Will receive guidance and perform a pelvic physiotherapy protocol after the evaluation, without the real-time monitoring by the physical therapist
  Interventions: Other: Pelvic physiotherapy
- Face-to-face group (Active Comparator): Will receive guidelines and will perform a pelvic physiotherapy protocol oriented in person by the physical therapist.
  Interventions: Other: Pelvic physiotherapy

INTERVENTIONS:
Other: Pelvic physiotherapy — All groups will receive the same treatment for 12 weeks, which will include floor muscle training pelvic floor, urge suppression techniques, bladder training and behavioral therapy.

SUMMARY:
The goal of this randomized clinical trial is to compare the effectiveness of a pelvic floor rehabilitation program in a face-to-face versus remote in community-dwelling elderly women with urinary incontinence. The main question it aims to answer is: What is the difference in effectiveness of a pelvic floor rehabilitation program through face-to-face versus remote intervention? Participants will be divided into three groups: Synchronous Group: will receive guidance and perform a real-time guided pelvic physiotherapy protocol through online physiotherapy by the physiotherapist, Asynchronous Group: will receive guidance and perform a pelvic physiotherapy protocol after the evaluation, without the real-time monitoring by the physical therapist and face-to-face group: will receive guidelines and will perform a pelvic physiotherapy protocol oriented in person by the physical therapist. All groups will receive the same treatment for 12 weeks, which will include floor muscle training pelvic floor, urge suppression techniques, bladder training and behavioral therapy. Participants will be evaluated pre-treatment, at the end of the 6th week, and at the end of 12 weeks.

DETAILED DESCRIPTION:
Aging is associated with changes in body composition, including a decrease in skeletal muscle mass. As a result, approximately 30-40% of the elderly may experience urinary incontinence, considered one of the most important geriatric syndromes, associated with a negative impact on quality of life. In clinical practice, pelvic floor muscle training and behavioral therapy promote positive effects on pelvic floor rehabilitation when performed and guided through face-to-face consultations. Through Telehealth, the aspects that refer to the role of the physiotherapist, technologies used and format of the approach do not seem to be clarified. Virtual home care is an accepted reality because it improves access to health care and has a positive effect on outcomes. However, barriers to its use can affect the accessibility. According to the World Health Organization, the definition of telehealth is "the provision of health services, where distance is a critical factor, by all health professionals, using information and communication technologies to exchange valid information for diagnosis, treatment and prevention of disease and injury, research and evaluation, and for the continuing education of health professionals, all in the interest of promoting the health of individuals and their communities". The World Confederation for Physical Therapy defines digital practice, "a term used to describe health services, support, and information provided remotely through digital communication and devices." The main objective is "to facilitate the effective delivery of Physical Therapy services, improving access to care and information, and managing health resources". In Brazil, the Federal Council of Physiotherapy and Occupational Therapy published the resolution for the practice of telehealth in a pandemic period, teleconsultation, telemonitoring and teleconsultation. Our hypothesis is that the synchronous and asynchronous communication between the physiotherapist and the participants, with or without the help of caregivers, may enable adherence to the home rehabilitation process when compared to face-to-face treatment, minimizing the effects of urinary incontinence. This study proposes to contribute to knowledge in the field of Pelvic Physiotherapy, in particular, through telehealth to provide the service of rehabilitation for elderly women with pelvic floor disorders, using the advancement of technology as a facilitator of synchronous and asynchronous communication, to approach elderly urinary incontinence and still compare the two forms of rehabilitation through telehealth with the face-to-face treatment. It is widely known that urinary incontinence is a factor of social inhibition for causing embarrassment, in addition to producing disturbance in the sleep in the face of increased nocturnal voiding frequency, directly affecting the quality of life of the elderly. The proposed safe and guided by a physiotherapist through three rehabilitation programs, synchronous telerehabilitation (in real time), asynchronous telerehabilitation (without real-time contact) and face-to-face rehabilitation, can be used to provide interventions in order to optimize health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or more;
* Urinary Incontinence for at least 12 months
* Internet access.

Exclusion Criteria:

* Pelvic cancer;
* Sling surgery;
* Urinary catheter;
* Antimuscarinic medication;
* Alzheimer;
* Parkinson;
* Multiple Sclerosis;
* Uncontrolled diabetes.

Ages: 60 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Presence of Urinary Incontinence. | Pre-treatment, at the end of the 6th week, at the end of 12 weeks.
  Application of The International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF)
Type of Urinary Incontinence. | Pre-treatment, at the end of the 6th week, at the end of 12 weeks.
  Type of UI by self-report question: What kind of Has leakage occurred more frequently in the last 7 days?
Frequency of Urinary Incontinence | Pre-treatment, at the end of the 6th week, at the end of 12 weeks.
  Self-reported frequency of leakage
Frequency of Urinary Incontinence. | Pre-treatment, at the end of the 6th week, at the end of 12 weeks.
  Self-reported use of pads.
Overactive bladder symptoms. | Pre-treatment, at the end of the 6th week, at the end of 12 weeks.
  Application of The International Consultation on Incontinence Questionnaire Overactive Bladder (ICIQ OAB)
Quality of Life. | Pre-treatment, at the end of the 6th week, at the end of 12 weeks.
  Application of The International Consultation on Incontinence Modular Questionnaire Lower Urinary Tract Symptoms Quality of Life (ICIQ- LUTSqol).

SECONDARY OUTCOMES:
Adherence to the study. | At the end of the 6th week and at the end of 12 weeks.
  Self-reported adherence to the protocol:
  Patients will report how many days they performed the guided exercises.
Patient's Satisfaction. | At the end of 12 weeks.
  Application of The MedRisk Instrument for Measuring Patient Satisfaction With Physical Therapy Care (MRPS).
Patient's Satisfaction. | At the end of 12 weeks.
  Application of The TELEHEALTH USABILITY QUESTIONNAIRE (TUQ)

CONTACTS AND LOCATIONS:
Overall Officials: Luís H. Telles da Rosa, Study Director — Federal University of Health Sciences of Porto Alegre (UFCSPA)
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altermann CD, Martins AS, Carpes FP, Mello-Carpes PB. Influence of mental practice and movement observation on motor memory, cognitive function and motor performance in the elderly. Braz J Phys Ther. 2014 Mar-Apr;18(2):201-9. doi: 10.1590/s1413-35552012005000150. PMID 24839046
- [Background] BØ, K. et al. Evidence-Based Physical Therapy for the Pelvic Floor: Bridging Science and Clinical Practice. 2. ed. London: Churchill Livingstone, 2015. E-book.
- [Background] Bradley CS, Brown JS, Van Den Eeden SK, Schembri M, Ragins A, Thom DH. Urinary incontinence self-report questions: reproducibility and agreement with bladder diary. Int Urogynecol J. 2011 Dec;22(12):1565-71. doi: 10.1007/s00192-011-1503-3. Epub 2011 Jul 28. PMID 21796472
- [Background] Brucki SM, Nitrini R, Caramelli P, Bertolucci PH, Okamoto IH. [Suggestions for utilization of the mini-mental state examination in Brazil]. Arq Neuropsiquiatr. 2003 Sep;61(3B):777-81. doi: 10.1590/s0004-282x2003000500014. Epub 2003 Oct 28. Portuguese. PMID 14595482
- [Background] da Mata KRU, Costa RCM, Carbone EDSM, Gimenez MM, Bortolini MAT, Castro RA, Fitz FF. Telehealth in the rehabilitation of female pelvic floor dysfunction: a systematic literature review. Int Urogynecol J. 2021 Feb;32(2):249-259. doi: 10.1007/s00192-020-04588-8. Epub 2020 Nov 11. PMID 33175229
- [Background] Dumoulin C, Morin M, Mayrand MH, Tousignant M, Abrahamowicz M. Group physiotherapy compared to individual physiotherapy to treat urinary incontinence in aging women: study protocol for a randomized controlled trial. Trials. 2017 Nov 16;18(1):544. doi: 10.1186/s13063-017-2261-4. PMID 29145873
- [Background] Engberg S, Sereika SM. Effectiveness of Pelvic Floor Muscle Training for Urinary Incontinence: Comparison Within and Between Nonhomebound and Homebound Older Adults. J Wound Ostomy Continence Nurs. 2016 May-Jun;43(3):291-300. doi: 10.1097/WON.0000000000000227. PMID 27163683
- [Background] INTERNATIONAL CONTINENCE SOCIETY. International Continence Society fact sheets. [S. l.], n. August, p. 1-40, 2015.
- [Background] Kang HG, Mahoney DF, Hoenig H, Hirth VA, Bonato P, Hajjar I, Lipsitz LA; Center for Integration of Medicine and Innovative Technology Working Group on Advanced Approaches to Physiologic Monitoring for the Aged. In situ monitoring of health in older adults: technologies and issues. J Am Geriatr Soc. 2010 Aug;58(8):1579-86. doi: 10.1111/j.1532-5415.2010.02959.x. Epub 2010 Jul 14. PMID 20646105
- [Background] Kincade JE, Dougherty MC, Carlson JR, Hunter GS, Busby-Whitehead J. Randomized clinical trial of efficacy of self-monitoring techniques to treat urinary incontinence in women. Neurourol Urodyn. 2007;26(4):507-511. doi: 10.1002/nau.20413. PMID 17366526
- [Background] LEE, Alan et al. Report of the Wcpt / Inptra Digital Physical Therapy Practice Task Force. [S. l.], n. May, p. 1-23, 2019.
- [Background] Pereira SB, Thiel Rdo R, Riccetto C, Silva JM, Pereira LC, Herrmann V, Palma P. [Validation of the International Consultation on Incontinence Questionnaire Overactive Bladder (ICIQ-OAB) for Portuguese]. Rev Bras Ginecol Obstet. 2010 Jun;32(6):273-8. doi: 10.1590/s0100-72032010000600004. Portuguese. PMID 20945012
- [Background] Poli-Neto OB, Chama PP, Romao AP, Dantas RA, Rosa-E-Silva JC, Candido-Dos-Reis FJ, Nogueira AA. Cultural Adaptation of the Patient Satisfaction Questionnaire and Validation of Its Use in the Portuguese Language for Women with Chronic Pelvic Pain. Rev Bras Ginecol Obstet. 2016 Sep;38(9):443-449. doi: 10.1055/s-0036-1592344. Epub 2016 Sep 19. PMID 27643519
- [Background] QUEIROZ, NEILA ALVES DE. TRADUÇÃO E ADAPTAÇÃO CULTURAL DO INTERNATIONAL CONSULTATION ON INCONTINENCE QUESTIONNAIRE FEMALE LOWER URINARY TRACT SYMPTOMS (ICIQ-FLUTS). [S. l.], p. 2, 2016.
- [Background] Rasche P, Wille M, Brohl C, Theis S, Schafer K, Knobe M, Mertens A. Prevalence of Health App Use Among Older Adults in Germany: National Survey. JMIR Mhealth Uhealth. 2018 Jan 23;6(1):e26. doi: 10.2196/mhealth.8619. PMID 29362211
- [Background] Tamanini JT, Dambros M, D'Ancona CA, Palma PC, Rodrigues Netto N Jr. [Validation of the "International Consultation on Incontinence Questionnaire -- Short Form" (ICIQ-SF) for Portuguese]. Rev Saude Publica. 2004 Jun;38(3):438-44. doi: 10.1590/s0034-89102004000300015. Epub 2004 Jul 8. Portuguese. PMID 15243675
- [Background] Virtuoso JF, Menezes EC, Mazo GZ. Effect of Weight Training with Pelvic Floor Muscle Training in Elderly Women with Urinary Incontinence. Res Q Exerc Sport. 2019 Jun;90(2):141-150. doi: 10.1080/02701367.2019.1571674. Epub 2019 Apr 4. PMID 30945991
- [Background] Ware P, Bartlett SJ, Pare G, Symeonidis I, Tannenbaum C, Bartlett G, Poissant L, Ahmed S. Using eHealth Technologies: Interests, Preferences, and Concerns of Older Adults. Interact J Med Res. 2017 Mar 23;6(1):e3. doi: 10.2196/ijmr.4447. PMID 28336506
- [Background] WHO. Telemedicine: opportunities and developments in Member States: report on the second global survey on eHealth 2009. Global Observatory for eHealth Series, [S. l.], v. 18, n. 2, p. 153, 2010.
- [Background] WORLD CONFEDERATION FOR PHYSICAL THERAPY. Digital Practice White Paper: Follow Up Survey. In: 2020, Anais [...]. [S. l.: s. n.]
- [Background] Yoon H, Jang Y, Vaughan PW, Garcia M. Older Adults' Internet Use for Health Information: Digital Divide by Race/Ethnicity and Socioeconomic Status. J Appl Gerontol. 2020 Jan;39(1):105-110. doi: 10.1177/0733464818770772. Epub 2018 Apr 16. PMID 29661052
- See also: Federal Council of Physiotherapy and Occupational Therapy resolution about the practice of telehealth — https://www.coffito.gov.br/nsite/?p=15825